CLINICAL TRIAL: NCT01266486
Title: A Phase 2 Single Arm Study to Examine the Effects of Metformin on Cancer Metabolism in Patients With Early Stage Breast Cancer Receiving Neoadjuvant Chemotherapy
Brief Title: Effect of Metformin on Breast Cancer Metabolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, Linda Ward, QA Coordinator, Cancer Centre, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EP-TSC-647
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Pharmacodynamics; AMPK; PET Scan
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Extended release Metformin 1500mg once daily for 14-21 days
  Other Names: Glucophage XR

SUMMARY:
Metformin, a drug that has been used since the 1950's in the treatment of diabetes, has recently generated great interest in its anticancer effects based on in vitro, in vivo and clinical studies. This study assesses the pharmacodynamic effects of metformin on breast cancer metabolism.

The trial design is based on a 2 centre study 'Early Antiangiogenic Response to Bevacizumab in Primary Breast Cancer' that is about to successfully complete recruitment in Oxford and Mount Vernon hospitals. The study takes advantage of the 2 week window between the first clinic visit and commencement of neoadjuvant chemotherapy. Metformin will be given to patients for at least 2 weeks prior to neoadjuvant chemotherapy with a set of 3 breast core biopsies, a PET-CT scan and blood tests carried out before and after this 2 week period of treatment. Patients will also receive a drink of heavy (deuterated) water, a safe and stable isotope commonly used in clinical lipid metabolism studies, the evening prior to both sets of core biopsies. Having completed the first 2 weeks of metformin patients will have the option of continuing metformin until completion of chemotherapy, at the discretion of the trial physician.

The core biopsies will then be used to assess for changes in:

* immunohistochemical staining;
* gene profiles;
* uptake of heavy water into tumour fatty acids using mass spectrometry techniques.

The aim is to identify potential biomarkers of response to metformin (and other future cancer metabolism drugs).

DETAILED DESCRIPTION:
Metformin is a safe and well tolerated drug that has been widely used in the treatment of diabetes for over 50 years. There is now growing evidence from in vitro laboratory and animal work that metformin has anticancer properties. In addition a retrospective clinical study in a diabetic population has demonstrated evidence of markedly increased pathological response rates (a typically robust surrogate clinical endpoint of efficacy) to pre-surgical chemotherapy in early breast cancer for patients that were also taking metformin as part of their diabetes treatment.

There are several studies of metformin in cancer patients ongoing or being developed worldwide These are predominantly in relatively unselected cancer populations and with clinical outcomes as endpoints. However this study is the only study currently planned which will carry out a substantial assessment of pharmacodynamic endpoints. It is important that this study is carried out at an early stage in the development of metformin as a potential cancer therapy in order to ensure that future large scale studies are properly informed.

ELIGIBILITY:
Inclusion Criteria:

* Women with histology proven locally advanced breast cancer (LABC) or tumours >3 cm in diameter.
* ECOG performance status 0-1.
* Age ≥18 years.
* No prior treatment for breast cancer and scheduled to commence neoadjuvant chemotherapy in <3 weeks time.
* Have given written informed consent and are capable of cooperating with protocol.
* Adequate bone marrow, renal and liver function.

Exclusion Criteria:

* Radiotherapy, major surgery, significant traumatic injury, endocrine therapy, immunotherapy, chemotherapy or experimental therapy during four weeks prior to starting or during trial.
* Pregnancy or breast feeding
* History of type 1 or type 2 diabetes.
* Serum glucose greater than 7.0 mMol/L.
* Treatment with metformin in the past year.
* Estimated glomerular filtration rate (eGFR) <45ml/min.
* Acute or chronic metabolic acidosis
* Known hypersensitivity to metformin
* Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Measure Metformin Induced effects in phosphorylation of S6K, 4E-BP-1 and AMPK via immunohistochemical analysis | after 14-21 days of daily metforming dosing

SECONDARY OUTCOMES:
Measure fatty acid desaturation and deuterated water uptake into fatty acids at baseline and after 2 weeks of metformin. | Day 14-21 after starting metformin dosing
Measure baseline and induced effect of metformin on upstream and downstream members of AMPK family via gene array analysis. | 14-21 days after start daily metformin dosing

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Harris, Principal Investigator — The University of Oxford
Locations (3):
- United Kingdom (3):
  - Mount Vernon Centre for Cancer Treatment, Rickmansworth Road, Northwood, Middlesex
  - Dept Oncology, Churchill Hospital, Old Road, Headington, Oxford, Oxfordshire
  - Surgery and Molecular Oncology Ninewells Hospital, Dundee, Scotland

REFERENCES:
- [Derived] Ralli GP, Carter RD, McGowan DR, Cheng WC, Liu D, Teoh EJ, Patel N, Gleeson F, Harris AL, Lord SR, Buffa FM, Fenwick JD. Radiogenomic analysis of primary breast cancer reveals [18F]-fluorodeoxglucose dynamic flux-constants are positively associated with immune pathways and outperform static uptake measures in associating with glucose metabolism. Breast Cancer Res. 2022 May 17;24(1):34. doi: 10.1186/s13058-022-01529-9. PMID 35581637
- [Derived] Lord SR, Collins JM, Cheng WC, Haider S, Wigfield S, Gaude E, Fielding BA, Pinnick KE, Harjes U, Segaran A, Jha P, Hoefler G, Pollak MN, Thompson AM, Roy PG, English R, Adams RF, Frezza C, Buffa FM, Karpe F, Harris AL. Transcriptomic analysis of human primary breast cancer identifies fatty acid oxidation as a target for metformin. Br J Cancer. 2020 Jan;122(2):258-265. doi: 10.1038/s41416-019-0665-5. Epub 2019 Dec 10. PMID 31819193
- [Derived] Lord SR, Cheng WC, Liu D, Gaude E, Haider S, Metcalf T, Patel N, Teoh EJ, Gleeson F, Bradley K, Wigfield S, Zois C, McGowan DR, Ah-See ML, Thompson AM, Sharma A, Bidaut L, Pollak M, Roy PG, Karpe F, James T, English R, Adams RF, Campo L, Ayers L, Snell C, Roxanis I, Frezza C, Fenwick JD, Buffa FM, Harris AL. Integrated Pharmacodynamic Analysis Identifies Two Metabolic Adaption Pathways to Metformin in Breast Cancer. Cell Metab. 2018 Nov 6;28(5):679-688.e4. doi: 10.1016/j.cmet.2018.08.021. Epub 2018 Sep 20. PMID 30244975